CLINICAL TRIAL: NCT06902896
Title: Safety and Efficacy of Immunosuppressive CAR-DC Targeting FAP in the Treatment of End-stage Dilated Cardiomyopathy
Brief Title: Safety and Efficacy of FAP iCDC in End-stage Dilated Cardiomyopathy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YAN2024-1210
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Dilated Cardiomyopathy (DCM); Heart Failure
Keywords: end-stage dilated cardiomyopathy; FAP immunosuppressive CAR-DC
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dilated cardiomyopathy (Experimental): Administration of FAP immunosuppressive CAR-DC cell therapy in dilated cardiomyopathy.
  Patients are planned to be enrolled in the dose-escalation trial (1×10^5/kg、4×10^5/kg、and 8×10^5/kg) .The first dose group (4×10⁵/kg) initially enrolls 3 subjects to observe Dose-Limiting Toxicity (DLT) responses.
  1. If no DLT occurs and all 3 subjects demonstrate efficacy after 6 months of treatment, and this dose is determined as the safe and effective dose.
  2. If 1 subject experiences DLT, 3 additional subjects are enrolled.
     * If 1/6 subjects develops DLT, and efficacy is not fully achieved in all 6 subjects, escalate to the next dose group (8×10^5/kg).
     * If ≥2/6 subjects develop DLT, de-escalate to the previous dose group (1×10^5/kg).
  Interventions: Biological: FAP immunosuppressive CAR-DC

INTERVENTIONS:
Biological: FAP immunosuppressive CAR-DC — Each subject receive FAP immunosuppressive CAR-DC by intravenous infusion

SUMMARY:
To study the safety and efficacy of fibroblast activation protein (FAP)-targeted immunosuppressive chimeric antigen receptor-dendritic cell (CAR-DC) in the treatment of end-stage dilated cardiomyopathy and provide a new method for the treatment of end-stage dilated cardiomyopathy.

DETAILED DESCRIPTION:
Background: Immune system activation and myocardial fibrosis are widely observed in patients with heart failure, whether it is ischemic or non-ischemic heart failure. Therefore, targeting inflammation and cardiac fibrosis may become a universal therapeutic strategy for the treatment of heart failure. At present, T cell surface molecular group modification (such as CAR-T) has been found to reduce fibrosis and restore cardiac function after injury in rodent heart failure models, suggesting that immune cells may be one of the potential effective targets for the treatment of heart failure. Dendritic cells (DCs) are the most powerful professional antigen-presenting cells in the body. Immature DCs have strong migration ability, and mature DCs can effectively activate naive T cells, which are at the center of initiating, regulating, and maintaining immune responses. Studies have confirmed that dendritic cells are involved in regulating inflammatory responses after myocardial injury.

Here, we innovatively applied chimeric antigen receptor (CAR) technology to edit DCs, making the new CAR immune cells exhibit an immunosuppressive phenotype, leading to T cell tolerance to CAR immune cells without producing new antigens; and targeting fibroblast activation protein (FAP) to accumulate in the fibrotic area of cardiac injury, thereby reducing fibrosis and enhancing cardiac function.

Purpose: To evaluate the efficacy and safety of immunosuppressive CAR-DC (iCDC) in the treatment of patients with end-stage dilated cardiomyopathy.

Study design: This study is a prospective, single-center, single-arm clinical study. The study objects are patients aged 18 to 75 years with end-stage dilated cardiomyopathy (ejection fraction < 35%) who visited the Department of Cardiology. In this study, patients with end-stage dilated cardiomyopathy were proposed to undergo FAP iCDC Cell therapy.

Outcome measure: The primary outcome is evaluation of the safety of FAP iCDC for end-stage dilated cardiomyopathy. The secondary outcomes are left ventricular ejection fraction (LVEF) assessed by echocardiography and cardiac magnetic resonance, enhanced volume assessed by cardiac magnetic resonance, interagency registry for mechanically assisted circulatory support (INTERMACS) grade, left ventricular internal dimension in systole (LVIDs), left ventricular internal dimension in diastole (LVIDd), left ventricular end-systolic volume (LVESV), left ventricular end-diastolic volume (LVEDV), N-terminal prohormone of brain natriuretic peptide (NT pro-BNP), 6 minutes walk test (6-MWT), New York Heart Association (NYHA) classification, Kansas City Cardiomyopathy Questionnaire (KCCQ) score, incidence of major adverse cardiac events (MACE) and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years old and 75 years old, diagnosed with dilated cardiomyopathy.
* Able to verbally confirm that he/she understands the risks, benefits and treatment options of the iCDC trial. He/she or his/her legal representative provides written informed consent before participating in the clinical trial.
* Diagnosed with Heart Failure with reduced ejection fraction (HFrEF), optimized drug therapy (under maximum tolerance of GDMT) for at least 3 months, left ventricular ejection fraction <35%, NYHA functional class ⅢB-IV, INTERMACS class 3-6.
* Blood test: hematocrit >30%, lymphocytes >0.5×10^9/L, platelets >60×10^9/L.

Exclusion Criteria:

* History of myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks before enrollment.
* CRT implanted within 12 weeks before enrollment or intended to implant CRT device.
* Previous heart transplantation or implantation of a ventricular assist device or similar device, or planned implantation of a ventricular assist device or similar device.
* Heart failure caused by ischemic cardiomyopathy, restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy, long-standing hypertension, congenital structural heart disease, or uncorrected primary valvular disease.
* Symptomatic bradycardia or second/third degree heart block.
* Active autoimmune disease requiring immunosuppressive therapy.
* Pulmonary Embolism (PE), Deep Vein Thrombosis(DVT), or recurrent embolism.
* A history of tuberculosis.
* History of severe renal failure or need for dialysis, creatinine >2.5 mg/dl.
* Uncorrected thrombocytopenia or systemic coagulopathy (platelet count < 50,000, INR > 2.5, or aPTT > 2.5 times control in the absence of anticoagulation), or active bleeding and uncorrectable coagulopathy.
* Aspartate aminotransferase or alanine aminotransferase levels greater than 5.0 times the upper limit of normal (ULN), total bilirubin >3 mg/dl.
* Systolic blood pressure <90 mmHg.
* History of concurrent severe infection, hepatobiliary obstruction, or malignancy.
* Infections: Active hepatitis B (PCR-detected hepatitis B virus DNA copies > 1000), hepatitis C, syphilis, or human immunodeficiency virus (HIV) infection at screening; uncontrolled systemic fungal, bacterial, viral, or other pathogen infection.
* Severe hemodynamic instability (eg, shock).
* Women who are pregnant or may become pregnant.
* Contraindications to study drugs or tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with Dose-limiting toxicity (DLT) | in 14 days after injection
  The proportion of participants with treatment-related adverse events as assessed by CTCAE v5.0
Incidence of treatment-emergent adverse events (TEAEs) | in 14 days after injection
  Incidence of iCDC treatment-emergent adverse events

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 1, 3, 6 months after injection
  The difference of LVEF from baseline. LVEF will be assessed by echocardiography.
Left ventricular ejection fraction (LVEF) | 6 months after injection
  The difference of LVEF from baseline. LVEF will be assessed by Cardiac Magnetic Resonance (CMR).
Enhanced volume (volume%) | 6 months after injection
  The difference of Enhanced volume (volume%) from baseline. Enhanced volume will be assessed by CMR.
INTERMACS Profile | 1, 3, 6 months after injection
  Profile 1. Critical cardiogenic shock; Profile 2. Progressive decline on inotropic support; Profile 3. Stable but inotrope dependent; Profile 4. Resting symptoms home on oral therapy; Profile 5. Exertion Intolerant; Profile 6. Exertion Limited; Profile 7. Advanced NYHA Class III symptoms
Left ventricular internal diameter end systole (LVIDs) | 1, 3, 6 months after injection
  The difference of LVIDs from baseline. LVIDs will be assessed by echocardiography.
Left ventricular internal diameter end diastole (LVIDd) | 1, 3, 6 months after injection
  The difference of LVIDd from baseline. LVIDd will be assessed by echocardiography.
Left ventricular end-systolic volume (LVESV) | 6 months after injection
  The difference of LVESV from baseline. LVESV will be assessed by CMR.
Left ventricular end-diastolic volume (LVEDV) | 6 months after injection
  The difference of LVEDV from baseline. LVEDV will be assessed by CMR.
NT-proBNP | 1, 3, 6 months after injection
  Analysis of differences of NT-proBNP serum level from baseline.
6 minutes walk test (6MWT) | 1, 3, 6 months after injection
  The difference of 6MWT from baseline.
assessment of heart failure symptom | 1, 3, 6 months after injection
  The difference of heart failure symptom, which will be assessed by NYHA grading and KCCQ score.
Incidence of major adverse cardiovascular events (MACE) | 1, 3, 6 months after injection
  Incidence of Cardiac death, readmission due to heart failure.
incidence of adverse events | 6 months
  Incidence of adverse events of heart, nerve system, mental system, digestive system and immune system.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang Hu, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No